CLINICAL TRIAL: NCT05744960
Title: The Impact of Clinic-level Financial Incentives on HPV Vaccine Communication and Uptake
Brief Title: Impact of Financial Incentives
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IMPACTP2FI; 1P01CA250989-01A1 (NIH)
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Human Papilloma Virus
Keywords: financial incentives; pediatric medicine; vaccination; pay-for-performance

STUDY DESIGN:
Intervention Model Description: Cluster randomized design in which clinics will be randomized within healthcare systems
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV vaccine communication training. (Experimental): Staff in clinics randomized to this arm will receive an intervention called Announcement Approach Training (AAT). This training is designed to improve communication about HPV vaccination.
  Interventions: Behavioral: Communication training
- HPV vaccine communication training and clinic-level financial incentive program (Experimental): Staff in clinics randomized to this arm will receive the Announcement Approach Training and a clinic-level financial incentive program with a monthly data feedback report to increase HPV vaccine uptake.
  Interventions: Behavioral: Communication training; Behavioral: financial Incentive

INTERVENTIONS:
Behavioral: Communication training — Clinics will host an Announcement Approach Training (AAT) workshop. A trained facilitator will use a standard script and slides to deliver workshop in-person or over Zoom; clinical staff who are unavailable will take the workshop later on their own.
Behavioral: financial Incentive — Clinics will host an AAT workshop, as in the other trial arm. Clinics in the intervention arm will then receive a 12-month clinic-level financial incentive program with predetermined targets for HPV vaccine initiation rates (5%, 10%, and 30% increases from baseline). Clinics will be notified of their HPV vaccination rates though a monthly, automated report. Clinic achievement will be assessed and incentives will be paid out to clinics monthly. Incentives will be tiered based on target and sized based on the number of clinic providers. For reaching the highest tier of 30%, clinics will receive an aggregate of $1000 per provider.
  Arms: HPV vaccine communication training and clinic-level financial incentive program

SUMMARY:
This trial will look at the impact of clinic-level financial incentives to improve provider communication and increase HPV vaccine uptake. Some clinics will receive communication training. Other clinics will receive the same training and a clinic-level financial incentive program with a monthly data feedback report to increase HPV vaccine uptake.

DETAILED DESCRIPTION:
The researchers will conduct a cluster randomized control trial. This trial will look at the impact of clinic-level financial incentives to improve provider communication and increase HPV vaccine uptake. The recruitment goal for the trial is 34 clinics in healthcare systems, including 9 rural-serving clinics. The researchers will randomize clinics using simple randomization (1:1). Some clinics will receive communication training. Other clinics will receive the same training and a clinic-level financial incentive program with a monthly data feedback report to increase HPV vaccine uptake. The researchers will use medical record data to compare changes in HPV vaccination among children ages 9-12. Clinics will be followed for 24 months. The study will engage clinical staff. Researchers will not have direct contact with children or their families.

ELIGIBILITY:
This trial will enroll clinics and intervene with clinical staff. We will use vaccination data from children to evaluate intervention effectiveness. We will not enroll children or interact with them directly.

Inclusion Criteria:

Clinics are eligible if they are a pediatric or family medicine clinic in North Carolina that in the past year had:

* less than 72% HPV vaccine initiation rate,
* greater than or equal to 50 patients ages 9-12
* greater than or equal to 2 HPV vaccine providers
* no clinic or provider-level financial incentive programs to increase system, clinic, or provider HPV vaccination rates among patients aged 9-12 in the past two years, and
* no HPV vaccine provider communication trainings in the past six months.

Children's medical records will be eligible to be included in the dataset if children:

* are between the ages of 9-12 years at baseline and
* are attributed to a participating clinic at 12- or 24-month follow-up.

Exclusion Criteria:

Clinics are excluded if they:

* do not provide HPV vaccine to children ages 9-12
* have a specialty other than pediatrics or family medicine
* had an HPV vaccine-specific financial incentive program in the past two years
* had a formal HPV vaccine communication training in the past 6 months
* had an HPV initiation rate greater than 72$
* had fewer than 49 patients aged 9-12
* had 1 or fewer HPV vaccine providers

Children's medical records will not be eligible to be included in the dataset if children:

* are not between the ages of 9-12 years at baseline
* are not attributed to a participating clinic at 12- or 24-month follow-up

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
HPV vaccination (≥1 dose), 9-12 year olds | from baseline to 12 months
  Proportion of unvaccinated children who initiate the HPV vaccine series between baseline and 12-month follow-up, among those who were ages 9-12 at baseline.

SECONDARY OUTCOMES:
HPV vaccination (≥1 dose), 9-12 year olds | from 13 months to 24 months
  Proportion of unvaccinated children who initiate the HPV vaccine series between 13- and 24-month follow-up, among those who were ages 9-12 at 13 months.
HPV vaccination (≥2 doses), 9-12 year olds | from baseline to 12 months
  Proportion of unvaccinated children who complete the HPV vaccine series between baseline and 12-month follow-up, among those who were ages 9-12 at baseline.
HPV vaccination (≥2 doses), 9-12 year olds | from 13 months to 24 months
  Proportion of unvaccinated children who complete the HPV vaccine series between 13- and 24-month follow-up, among those who were ages 9-12 at 13 months.

CONTACTS AND LOCATIONS:
Overall Officials: Justin G Trogdon, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No